CLINICAL TRIAL: NCT05933889
Title: Single and Combined Modality Trans-Oral Robotic Surgery in Early Oropharyngeal Cancer: Exploring the Impact of Surgical Margins on Local Disease Recurrence: The SCORE Study
Brief Title: Single and Combined Modality Trans-Oral Robotic Surgery in Early Oropharyngeal Cancer
Acronym: SCORE
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5852; CCR5852 (Other: Royal Marsden Committee for Clinical Research); IRAS327707 (Other: UK NHS HRA)
Record Dates: First submitted 2023-06-14; First posted 2023-07-06 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Cancer Head Neck
Keywords: Robotic Surgical Procedures; Margins of Excision; Oropharyngeal neoplasms; Local neoplasm recurrence; Recurrence free survival
MeSH Terms: conditions — Head and Neck Neoplasms; Margins of Excision; Oropharyngeal Neoplasms; Neoplasm Recurrence, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Samples to be collected for germline and circulating tumour DNA analysis:
  * Blood
  * Buccal swabs
  Samples to be taken as part of standard care for molecular analysis:
  - Fresh or Archival Tumour tissue (biopsies and resections)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective observational cohort: Retrospective patients undergoing transoral robotic surgery for early stage T1-2 oropharyngeal cancers on or before to 31/12/2021. Data will be collected from medical records.
- Exploratory molecular analysis: Consenting prospective patients based in the UK identified will be invited to participate in the exploratory molecular analysis by their usual care team. If agreeable, patients will consent to donation of either blood or buccal swab samples, in addition to archival tissue from their primary, and if relevant, recurrent tissue samples.
  Interventions: Genetic: Molecular Analysis
- Radiology/ radiomic analysis: Retrospective patients based in the UK and abroad will have their pre-operative imaging transferred to the RMH radiology department which will undergo radiomic and morphological assessment to ascertain features that put patients at high risk of local recurrence and positive margins.
  Interventions: Other: Radiomic/ Morphological analysis

INTERVENTIONS:
Genetic: Molecular Analysis — Germline and circulating tumour DNA analysis of buccal/ blood samples and molecular analysis of primary and recurrent tumour tissue samples
  Groups: Exploratory molecular analysis
Other: Radiomic/ Morphological analysis — Radiomic analysis and assessment of morphological features of pre-operative CT/ MRI imaging in patients who have undergone TORS for primary oropharyngeal cancer.
  Groups: Radiology/ radiomic analysis

SUMMARY:
Multi-centre retrospective observational cohort study with optional exploratory radiomic study (international) and prospective molecular analysis studies (UK only).

DETAILED DESCRIPTION:
The SCORE study is a international multicentre cohort study investigating the local recurrence free survival outcomes in patients undergoing transoral robotic surgery with and without adjuvant therapy for early stage (T1-T2) oropharyngeal squamous cell carcinoma (OPSCC). Important secondary objectives include assessment of other survival measures (overall, disease free and disease specific), determination of a safe margin "cut off" that minimises the risk of local recurrence, and reporting the rate of early post-operative complications and mortality.

Retrospective SCORE patients will optionally contain an exploratory radiomic and radiology morphological analysis to ascertain high risk features of positive margins and local recurrence following TORS for early oropharyngeal cancer.

Additionally, the SCORE study will contain a prospective exploratory molecular analysis of consenting patients to help further define OPSCC molecular characteristics in those who experience recurrence and those who do not, in addition to assessing levels of circulating tumour DNA in before and after TORS procedures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older.
* Primary tumour within the oropharynx (defined as tonsil, soft palate, tongue base, lateral and posterior oropharyngeal walls)
* Histologically confirmed squamous cell carcinoma.
* P16 positive or negative tumours
* Index cancer treated with TORS with or without adjuvant therapy.
* Early pT1-T2 stage oropharyngeal SCC
* TORS performed on or before 31st December 2021

For the exploratory analysis only:

* Ability to consent to molecular analysis study
* Ability to consent to radiomic/ imaging study (as required for international centres)

Exclusion Criteria:

* Moderate to advanced stage T3-T4 oropharyngeal SCC
* TORS performed for diagnostic, recurrent, or palliative intentions.
* Prior history of head and neck cancer or radiation therapy at any time
* Known distant metastatic disease.
* Nasopharyngeal, thyroid, cutaneous, and non-SCC head and neck cancers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older diagnosed with early (T1-T2) primary oropharyngeal squamous cell carcinoma, treated with transoral robotic surgery with or without adjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
To report 2-year locoregional survival outcomes following TORS for primary OPSCC with or without adjuvant therapy | 2 years
  To report 2-year locoregional survival outcomes following TORS for primary OPSCC with or without adjuvant therapy

SECONDARY OUTCOMES:
To report 2-year overall survival outcomes following TORS for primary OPSCC with or without adjuvant therapy. | 2 years
  To report 2-year overall survival outcomes following TORS for primary OPSCC with or without adjuvant therapy.
To report 2-year disease-free survival outcomes following TORS for primary OPSCC with or without adjuvant therapy. | 2 years
  To report 2-year disease-free survival outcomes following TORS for primary OPSCC with or without adjuvant therapy.
To report 2-year disease specific survival outcomes following TORS for primary OPSCC with or without adjuvant therapy. | 2 years
  To report 2-year disease specific survival outcomes following TORS for primary OPSCC with or without adjuvant therapy.
Define the optimum margin cut off required to avoid 2-year locoregional recurrence in primary TORS without adjuvant therapy | 2 years
  Define the optimum margin cut off required to avoid 2-year locoregional recurrence in primary TORS without adjuvant therapy
To report rates of 30-day post-operative mortality | 30 days
  To report rates of 30-day post-operative mortality
To report rates of 30-day post-operative haemorrhage | 30 days
  To report rates of 30-day post-operative haemorrhage
To report rates of 30-day major haemorrhage necessitating surgical intervention | 30 days
  To report rates of 30-day major haemorrhage necessitating surgical intervention
To report long term feeding tube use after primary TORS surgery with and without post-operative radiotherapy | 12 months
  To report the rate of feeding tube use at 12 months post-operatively
To report long term tracheostomy tube use after primary TORS surgery with and without post-operative radiotherapy | 12 months
  To report the rate of tracheostomy tube use at 12 months post-operatively
Identify clinical and pathological factors predictive of 2-year survival outcomes on uni- and multivariate analysis | 2 years
  Identify clinical and pathological factors predictive of 2-year survival outcomes on uni- and multivariate analysis

OTHER OUTCOMES:
Ascertain the differing molecular characteristics between tumours that experience early 2-year local recurrence and those who do not. | 2 years
  Ascertain the differing molecular characteristics between tumours that experience early 2-year local recurrence and those who do not.
Ascertain the changes in circulating tumour DNA levels in patients undergoing primary TORS for early oropharyngeal cancer. | 2 years
  Ascertain the changes in circulating tumour DNA levels in patients undergoing primary TORS for early oropharyngeal cancer.
Correlation of high-risk genetic features with 2 year local recurrence outcomes | 2 years
  Correlation of high-risk genetic features with 2 year local recurrence outcomes
Ascertain CT or MRI radiomic/ or morphological characteristics of tumours that develop 2-year local recurrence. | 2 years
  Ascertain CT or MRI radiomic/ or morphological characteristics of tumours that develop 2-year local recurrence.
Correlation of high-risk radiomic/ or morphological features and local recurrence | 2 years
  Correlation of high-risk radiomic/ or morphological features and local recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Vinidh Paleri, Principal Investigator — Royal Marsden Hospital NHS Foundation Trust
Locations (1):
- The Royal Marsden Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hardman JC, Holsinger FC, Brady GC, Beharry A, Bonifer AT, D'Andrea G, Dabas SK, de Almeida JR, Duvvuri U, Floros P, Ghanem TA, Gorphe P, Gross ND, Hamilton D, Kurukulasuriya C, Larsen MHH, Lin DJ, Magnuson JS, Meulemans J, Miles BA, Moore EJ, Pantvaidya G, Roof S, Rubek N, Simon C, Subash A, Topf MC, Van Abel KM, Vander Poorten V, Walgama ES, Greenlay E, Potts L, Balaji A, Starmer HM, Stephen S, Roe J, Harrington K, Paleri V. Transoral Robotic Surgery for Recurrent Tumors of the Upper Aerodigestive Tract (RECUT): An International Cohort Study. J Natl Cancer Inst. 2022 Oct 6;114(10):1400-1409. doi: 10.1093/jnci/djac130. PMID 35944904
- [Background] Warner L, O'Hara JT, Lin DJ, Oozeer N, Fox H, Meikle D, Hamilton D, Iqbal MS, Robinson M, Paleri V. Transoral robotic surgery and neck dissection alone for head and neck squamous cell carcinoma: Influence of resection margins on oncological outcomes. Oral Oncol. 2022 Jul;130:105909. doi: 10.1016/j.oraloncology.2022.105909. Epub 2022 May 26. PMID 35636080
- [Background] Williamson A, Moen CM, Slim MAM, Warner L, O'Leary B, Paleri V. Transoral robotic surgery without adjuvant therapy: A systematic review and meta-analysis of the association between surgical margins and local recurrence. Oral Oncol. 2023 Dec;147:106610. doi: 10.1016/j.oraloncology.2023.106610. Epub 2023 Nov 9. PMID 37951118